CLINICAL TRIAL: NCT05887037
Title: Economic Impact of Metagenomic Next-generation Sequencing Versus Traditional Bacterial Culture Directed CNSIs Diagnosis and Therapy in Post-neurosurgical Patients Using a Decision Analysis Model
Brief Title: Economic Impact of mNGS on Diagnosis of Post-neurosurgical Central Nervous System Infection
Acronym: mNGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-018-02
Record Dates: First submitted 2023-05-07; First posted 2023-06-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Central Nervous System Infections
Keywords: Central nervous system infections; Metagenomic next-generation sequencing
MeSH Terms: conditions — Central Nervous System Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group was sent for CSF mNGS and traditional microbiological cultures at the same time, and the mNGS results were usually earlier than the traditional microbiological cultures results. The experimental group adjusted or continued the current medication regimen according to the mNGS reporting pathogen and the expert team's opinion. Subsequently, if the CSF traditional microbiological cultures results in the experimental group are consistent with the mNGS results, the current treatment plan of the patient is continued, and if the results are inconsistent with the mNGS results, the expert team needs to discuss and adjust the treatment plan. When no causative organism is detected in mNGS, empiric treatment is continued, and treatment is adjusted pending the pathogen culture results.
  Interventions: Diagnostic Test: mNGS; Diagnostic Test: The traditional microbiological cultures
- Control group (Active Comparator): After a clinical diagnosis of central nervous system infection, the control group was treated empirically based on only cerebrospinal fluid for traditional microbiological cultures, without mNGS detection, and the treatment plan was adjusted according to the traditional microbiological cultures results. If the patient's culture is negative and empiric therapy does not improve, cerebrospinal fluid is retained for mNGS testing. Treatment is adjusted based on mNGS results and expert team evaluation.
  Interventions: Diagnostic Test: The traditional microbiological cultures

INTERVENTIONS:
Diagnostic Test: mNGS — mNGS is the direct extraction of nucleic acid from clinical samples. High-throughput sequencing technology and bioinformatics analysis were adopted to complete the detection of pathogens such as bacteria, fungi, viruses and parasites at one time
  Arms: Experimental group
Diagnostic Test: The traditional microbiological cultures — Traditional microbial culture is the gold standard for the diagnosis of central nervous system infection, but the traditional microbiological culture time is long and the detection rate is low.

SUMMARY:
The aim of the current study was to assess the economic impact of using metagenomic next-generation sequencing (mNGS) versus traditional bacterial culture directed CNSIs diagnosis and therapy in post-neurosurgical patients from Beijing Tiantan Hospital. mNGS is a relatively expensive test item, and whether it has the corresponding health economic significance in the clinical application of diagnosing intracranial infection has not been studied clearly. Therefore, the investigators hope to explore the clinical application value of mNGS detection in central nervous system infection after neurosurgery.

DETAILED DESCRIPTION:
Central nervous system infections (CNSIs) are severe complications after neurosurgery, that can lead to a poor prognosis. The incidence of postoperative central nervous system infections (PCNSIs) ranges from 2.8% to 14%, and there are differences between different regions. The incidence rate in developed countries is lower than that in developing countries. The most common manifestations of PCNSIs include meningitis, ventriculitis, subdural abscess, epidural abscesses, and brain abscesses. Studies have shown that the most common pathogens of PCNSIs are Staphylococcus aureus, and coagulase-negative staphylococcus, followed by gram-negative bacteria. In China, the pathogen detection rate of traditional cerebrospinal fluid (CSF) culture can only reach 5.4-10%. In addition, culture as the gold standard is time-consuming and susceptible to the use of antibiotics. PCNSIs is related to increased treatment costs, prolonged hospitalization time, psychological trauma and delayed postoperative adjuvant treatment, which places a substantial economic and psychological burden on society and patients' families.

Given the seriousness of PCNSIs, it is challenging to choose the appropriate antibiotic treatment for PCNSIs and should be guided by pathogens and their drug sensitivity. Thus, early and efficient diagnosis of pathogens is crucial for PCNSIs. Compared with traditional pathogenic microbial detection methods, metagenomic next-generation sequencing (mNGS) has faster, more accurate, and more complete advantages. Currently, it is widely used in CNSIs, respiratory infections, blood infections, etc., especially suitable for the diagnosis of acute, critical, and complicated infections. Studies have shown that the positive rate of mNGS is much higher than that of culture, and it is less affected by the use of antibiotics, which can provide more accurate feedback on the patient's infection status. At the same time, it can detect a variety of pathogen types, providing more effective guidance for treatment. In addition, the fast detection speed of mNGS can effectively shorten the patient's course of the disease and significantly improve the prognosis of infected patients.

Most published mNGS studies are evaluations of their clinical diagnostic value. However, there is still some controversy over the full clinical use of mNGS, and one of the main reasons is cost constraints. The overall cost of mNGS detection reagents and labor in each sample is much higher than that of traditional detection methods. There are still no reports on health economics research on the use of mNGS to diagnose CNSIs after neurosurgery. Therefore, prospective clinical trials are needed to evaluate the cost-effectiveness of mNGS, a relatively expensive new detection method.

In summary, this study intends to conduct a health economics study of mNGS to diagnose postoperative central nervous system infections and evaluate whether mNGS, as a relatively expensive new technology, can identify the pathogen at the early stage, shorten the time of anti-infective treatment, reduce the overall medical cost, and improve the cure rate of patients. In addition, this study provides theoretical guidance for clinical and public health departments to make cost-effective decisions more scientifically, make more effective use of medical resources, and improve the social and economic benefits of etiological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

·Central nervous system infections

Exclusion Criteria:

* Unqualified samples
* Patients and their families refused to sign the informed consent
* The clinician considered the case unsuitable for inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Incremental cost effectiveness ratio | up to 12 weeks
  Measures the increased cost for each unit of mortality reduction or increase in cure rate

SECONDARY OUTCOMES:
Cost comparison | up to 12 weeks
  The difference in total cost between the mNGS group (experimental group) and the etiology culture group (control group) was compared, and the time cost, detection cost, anti-infection treatment-related cost and other costs were calculated respectively.
Efficacy comparison | up to 12 weeks
  The cure rate and mortality rate of central nervous system infection in the experimental group, and the control group were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Linlin Zhang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No